CLINICAL TRIAL: NCT00659971
Title: A Phase 2B Dose-Ranging Study of PAC113 Mouthrinse for Clinical and Microbial Evaluation in HIV Seropositive Individuals With Oral Candidiasis to Establish the Optimal Dose of PAC113
Brief Title: Phase 2B Dose-Ranging Study of PAC113 Mouthrinse in HIV Seropositive Individuals With Oral Candidiasis
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Pacgen Biopharmaceuticals Corporation (Industry)
Collaborators: Quintiles, Inc. (Industry)
Responsible Party: Pacgen Biopharmaceuticals Corp., Director, Drug Development
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: PBC002-01
Record Dates: First submitted 2008-03-18; First posted 2008-04-17 (Estimated); Last update posted 2008-06-26 (Estimated); Status verified 2008-06

CONDITIONS: Oral Candidiasis
Keywords: oral candidiasis
MeSH Terms: conditions — Candidiasis, Oral

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- 1 (Experimental): PAC113 0,15% mouthrinse
  Interventions: Drug: PAC113
- 2 (Experimental): PAC113 0,075% mouthrinse
  Interventions: Drug: PAC113
- 3 (Experimental): PAC113 0,0375% mouthrinse
  Interventions: Drug: PAC113
- 4 (Active Comparator): Nystatin suspension
  Interventions: Drug: PAC113

INTERVENTIONS:
Drug: PAC113 — PAC113 mouthrinse 0.15%; 0.075%; 0.0375% QID for 14 days

SUMMARY:
The purpose of this study is to determine the optimal dose of PAC113 mouthrinse for treatment of oral candidiasis in HIV seropositive patients.

DETAILED DESCRIPTION:
This is a randomized, examiner-blinded, positive-controlled, parallel design clinical trial, which features 4 treatment arms. Forty-five (45)* HIV positive subjects per treatment arm will be recruited for 180 subjects total. The study includes 5 visits: a screening visit, a 14-day treatment phase with a baseline visit on Day 1, a Day 7 visit, a post-treatment visit 5 days after the last dose, and follow-up visit. During the screening visit subjects will be assessed for study eligibility. Eligible subjects will be randomized to 1 of the following treatment arms:

A. 0.15% PAC-113 mouthrinse (5 mL 4 times daily [q.i.d.]); B. 0.075% PAC-113 mouthrinse (5 mL q.i.d.); C. 0.0375% PAC-113 mouthrinse (5 mL q.i.d.); D. Nystatin oral suspension (100,000 units/mL; 5 mL q.i.d.) Subjects will be evaluated clinically for safety and severity of clinical signs and symptoms of oral candidiasis at baseline (Day 1), Day 7, Day 19 (5 days post-treatment) and Day 28 (follow-up visit). Subjects will also have a microbiological analysis performed at screening, and at Days 7, 19 and 28.

ELIGIBILITY:
Inclusion Criteria:

* Are male or female 18 to 65 years of age, inclusive
* Are able and willing to follow study procedures and instructions
* Are able to read, understand and sign an informed consent form
* Are documented as HIV positive
* Have pseudomembranous and/or erythematous oral candidiasis as confirmed by potassium hydroxide preparation of mucosal scraping
* Have a CD4 cell count performed prior to randomization or within 6 weeks prior to the screening visit
* Have a viral load performed prior to randomization or within 6 weeks prior to the screening visit.
* Both men and women who are active heterosexually must be willing to practice a medically accepted method of birth control.

Exclusion Criteria:

* Have received systemic antifungal therapy within 14 days of starting study
* Have received prior topical therapy for oral candidiasis within 7 days of starting study
* Have a concomitant fungal infection requiring systemic therapy
* Are currently receiving immunosuppressive therapy (e.g. corticosteroids), or cancer chemotherapy
* Female subjects who are pregnant (as determined by a positive serum or urine pregnancy test) or lactating, or female subjects who are of childbearing potential and who are not using hormonal or barrier methods of birth control (e.g., oral or parenteral contraceptives, diaphragm plus spermicide, condoms) or who have not characterized themselves as abstinent. Subjects who use hormonal contraceptives must have started the method at least 30 days prior to the screening examination
* Active substance abuse
* Have esophageal symptoms (dysphagia or odynophagia) unless esophageal candidiasis has been ruled out by endoscopy
* Have a life expectancy < 4 weeks
* Are currently receiving or have received an investigational agent in the last 30 days
* Have had a change in antiretroviral therapy within 14 days prior to study entry (this does not apply to dose adjustment of the same therapy)
* Have any of the following laboratory abnormalities:

  * White blood cell (WBC) count <1,500 cells/mm3
  * Neutrophil granulocyte count <1,000 cells/mm3
  * Hemoglobin <9.0/dL
  * Transaminases (alanine aminotransferase [ALT] or aspartate aminotransferase [AST]) or bilirubin >3 times the upper limit of normal (ULN)
  * Serum creatinine >2 times ULN
* Have peri-oral lesion (perleche) only
* Have oral manifestations of herpes simplex (active disease only), hairy leukoplakia and/or aphthous ulcers

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 223 (Actual)
Dates: Start 2008-01; Primary Completion 2008-06 (Actual); Study Completion 2008-06 (Actual)

PRIMARY OUTCOMES:
Eliminating or reducing clinical signs and symptoms of oral Candida infections. | Day 19

SECONDARY OUTCOMES:
To evaluate the microbiological response of Candida to different concentrations of PAC-113. | Day 19

CONTACTS AND LOCATIONS:
Locations (1):
- Rosedale Infectious Disease, Huntersville, North Carolina, United States